CLINICAL TRIAL: NCT01177449
Title: The Effect of Prolotherapy on Balance and Lumbar Flexibility in the Patients With a Sacralized L5 Vertebra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Department of Rehabilitation Medicine, Chang Gung Medical Foundation, Linkou Branch, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-1825B
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Lumbosacral Transitional Vertebra
Keywords: prolotherapy
MeSH Terms: interventions — Prolotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Prolotherapy — inject normal saline and 50% glugose water with 1:1 ratial in volumn
  Other Names: Proliferative Injection Therapy

SUMMARY:
The purpose of this study is to investigate the effect of prolotherapy on balance and lumbar flexibility in the patients with a sacralized L5 vertebra. Evaluations for ability on balance include sensory organization test (SOT,) rhythmic weight shifting (RWS) and limits of stability (LOS.)

DETAILED DESCRIPTION:
Lumbosacral transitional vertebra (LSTV) is a congenital variety of vertebral bony construction, which is most frequently presented as sacralized L5 or lumbarized S1. LSTV would alter the kinetics of the spine thus induce inadequate mobility and dynamic compensation. Patients with LSTV were commonly found when they visited clinicians for treatment of low back pain. Prolotherapy is a technique that stimulates the body to repair the painful area by assistance of injecting an otherwise non-pharmacological and non-active irritant solution into the body.

ELIGIBILITY:
Inclusion Criteria:

* patients with a sacralized L5 vertebra confirmed by X-ray images

Exclusion Criteria:

* neuromuscular injury
* visual deficit
* vestibular deficit
* cannot recognize the marks on the screen

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
sensory organization | 30 minutes
rhythmic weight shifting | 30 minutes
limits of stability | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Wei Chou, MD, PhD., Principal Investigator — Department of Rehabilitation Medicine, Chang Gung Medical Foundation, Linkou Branch
Locations (1):
- Department of Rehabilitation Medicine, Chang Gung Medical Foundation, Linkou Branch, Guishan, Taoyuan County, Taiwan